CLINICAL TRIAL: NCT05412329
Title: Open- Label Phase I Study to Assess the RP2D of GC012F CAR-T in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Dual Targeted CD19/BCMA FASTCART GC012F in Relapsed/ Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Juan Du, Clinical Professor, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC012F-31
Record Dates: First submitted 2022-06-04; First posted 2022-06-09 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC012F treatment (Experimental): R/R multiple myeloma patients be treated with a single dose of GC012F cells.
  Interventions: Biological: GC012F injection

INTERVENTIONS:
Biological: GC012F injection — GC012F injection is a autologous dual CAR-T targeted BCMA and CD19. A single infusion of CART cells will be administered intravenously.

SUMMARY:
This is a single-arm, non-randomized, open-label study to confirm the RP2D (recommended phase 2 dose) of GC012F injection in patients with Relapsed/Refractory multiple myeloma (RRMM).

DETAILED DESCRIPTION:
This is a single-arm, non-randomized, open-label study to evaluate the RP2D of GC012F injection in patients with Relapsed/Refractory multiple myeloma (RRMM).

Approximately 6-9 eligible patients will be enrolled in escalating dosing cohorts to evaluate the RP2D of GC012F injection. Pts will be enrolled concurrently and assessed for ORR and DLT in respective dosing cohort. Based on this assessment the RP2D will be confirmed.

Table1 Dose Level Dose Level DL-1 DL1 DL2 Dose 1×105 /kg 2×105 /kg 3×105 /kg Patients who signed the informed consent will be screened for inclusion/exclusion criteria, and 3 eligible subjects will be enrolled in DL1.

1. After the DLT observation period of 21 days, if ≤1 of the first 3 subjects has a DLT event, 3 additional subjects will be enrolled in DL1.

   - ORR will be assessed at prespecified timepoints up to 24-weeks post treatment.

   A. If ORR > 66%, the study concludes and respective dose level will be determined as RP2D B. If ORR≤66%, 3 subjects will be enrolled in DL2
2. If > 1 of the 3 enrolled subjects has a DLT event, 3 more subjects will be enrolled in the lower dose level

2. During the DLT observation period, if > 1 of the first 3 subjects has a DLT event, 3 subjects will be enrolled in DL-1 to evaluate safety.

Patients in each dose group will be closely observed for at least 21 days post GCO12F infusion for DLT. Safety and DLT will be assessed by SMC according to definition of protocol for DLT. There will be no fixed dose interval between each dose level and each patient within the dose cohort. In addition, after one year of infusion, patients will be rolled over to a protocol for long-term safety to assess risk of RCL and lentivirus insert in vivo.

This study will be divided into six parts: screening, apheresis, baseline assessment, lymphodeleption, CAR-T cell infusion, and follow-up. Eligible patients will be apheresed and infused after CAR-T product release, patients will receive a 3-days standard F/C chemotherapy regimen for lymphodeleption. The recommend regimens for chemotherpay are as follows

FC regimen:

1. Fludarabine 30 mg/m2/d, iv gtt for 3 days;
2. Cyclophosphamide 300 mg/m2/d, iv for 3 days. GC012F infusion will be performed at 48-72 hours after chemotherapy pretreatment.

After GC012F infusion, subjects will be followed for safety and efficacy up to 1 year, or disease progression, death or withdrawal whichever comes earlier. In case of progression of disease,subsequent survival follow-up (survival state only) will be performed every 84 days (12 weeks) ± 14 days (2 weeks) till death,loss of follow up, or withdraw of consent. If there is no disease progression after 1 year of infusion, the same follow-up for survival will be carried out as mentioned above. End of this study will be 1 year after the last patient received infusion with GC012F.

All patients who complete the study, as well as those who discontinue from the study after receiving GC012F for reasons other than death, will be asked to participate in a 15 years follow-up study to monitor RCL and lentivirus insert sites in vivo.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients should meet all the following criteria:

1. Age of 18-70 years at the time of signing informed consent (contains critical values)；
2. Documented diagnosis at initial of active multiple myeloma according to IMWG criteria, and meet one or more of the following criteria at screening:

   1. Serum M protein ≥ 1 g/dL
   2. Urine M protein ≥ 200 mg/24h
   3. Serum free light chain sFLC ≥ 10 mg/dL with abnormal serum κ/λ ratio
3. Have had at least 3 different prior lines of therapy or primary refractory and PD within 12 months of their last line of therapy (patient should undergo at least 1 complete cycle of treatment in each line of therapy) defined by Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1; or patients have had at least 2 different prior lines of therapy and refractory to both IMiD and PI;
4. Estimated life expectancy ≥3 months;
5. ECOG: 0 or 1;
6. Hemoglobin ≥ 7.0 g/dL (without prior RBC transfusion within 7 days before screening; recombinant human erythropoietin use is permitted);
7. Absolute neutrophil count ≥ 1×109/L (without recombinant human granulocyte colony-stimulating factor within 7 days before screening and without pegylated G-CSF within 14 days of the laboratory test);
8. Platelet count ≥50×109/L(without prior platelet transfusion within 7 days before the laboratory test)
9. Absolute lymphocyte count ≥ 0.1×109/L;
10. Adequate functional reserve of organs:

    1. ALT/AST ≤ 2.5× UNL (upper normal limit);
    2. Serum creatinine > 45 mL/min, calculated by Cockcroft-Gault;
    3. Serum total bilirubin ≤ 2× UNL, except in subjects with congenital bilirubinemia (for participants with Gilbert syndrome, direct bilirubin ≤ 1.5× UNL is required);
    4. Calibrated serum calcium ≤ 12.5 mg/dL (≤ 3.1 mmol/L) or free ionized calcium ≤ 6.5 mg/dL (≤ 1.6 mmol/L);
11. Sufficient venous access for leukapheresis collection, and no other contraindications to leukapheresis;
12. Woman of childbearing age must have serum HCG negative during screen and baseline. Males agreed to avoid sperm donation at least 1 year after GC012F infusion. Males and sexual partner with fertility are willing to use effective and reliable method of contraception for at least 1 year after infusion;
13. Ability and willingness to adhere to the study visit schedule and all protocol requirements;
14. Subjects themselves or their legal representatives must voluntarily sign written informed consent form(s).

Exclusion Criteria:

• Patients should be excluded if they meet any one of the following criteria:

Exclusion criteria:

Patients should be excluded if they meet any one of the following criteria:

1. Presence of plasma cell leukemia (absolute number of peripheral plasma cells >2.0×109/L), Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein disease, skin changes) or primary amyloidosis (AL) at screening;
2. Patients have other aggressive malignancies (except patients with disease free survival for more than 5 years from non-melanoma skin cancer and cervical carcinoma in situ, bladder cancer, or breast cancer);
3. Any situations not benefit for subjects to accept or tolerated to planned therapy or understand informed consent; or any situation in which investigators believe that participation in this study is not in the subject's best interests (e.g., harm to health), or any situation that may prevent, limit or confuse the assessment;
4. Patients with prior history of seizures or stroke within 6 months before signing ICF;
5. Patients following cardic condition:

   1. New York Heart Association (NYHA) III or IV heart failure;
   2. Myocardial infarction or coronary artery bypass graft (CABG) ≤ 6 months prior to signing ICF;
   3. History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration;
   4. History of severe non-ischemic cardiomyopathy;
   5. Impaired cardiac function (left ventricular ejection fraction [LVEF] < 45%) as assessed by echocardiography or multiple gated acquisition scanning, or other heart diseases with clinically significant symptoms in 6 months prior to enrollment;
6. Patients have known active, or history of central nervous system involvement or exhibit clinical signs of meningeal involvement in multiple myeloma;
7. Patients positive for any of the following tests:

   1. HIV antibody;
   2. HCV antibody, those who are positive need to be tested for HCV-RNA, and those below the lower limit of the detection value can be enrolled;
   3. HBsAg or HBcAb; if HBcAb positive then HBV DNA copies will be further detected by PCR with machine of COBAS AmpliPrep/COBAS Taqman (or other methods with equal sensitivity) and result negative patients can be enrolled.
   4. TPPA antibody;
8. Suspect or evidence of serious active viral, bacterial or uncontrolled systemic fungal infections needs system anti-infection; active autoimmune disease or a history of autoimmune disease within 3 years prior to signing ICF;
9. Exist of pulmonary fibrosis;
10. Allergy subjects or history of severe hypersensitivity;
11. Oxygen inhalation requirement to maintain adequate oxygen saturation;
12. Patients have major surgery performed within 2 weeks prior to signing ICF, or planned during the study or within 2 weeks after GC012F infusion (except subjects who are planned for local anesthesia surgery);
13. Chemotherapy forbidden for cyclophosphamide and fludarabine;
14. Any tubes inserted or drain pipes except central venous catheter;
15. Pregnant or breast-feeding women who are and unwilling to stop breastfeeding, or men who are planned to have babies within 1 year of receiving treatment;
16. Patients who have received any prior therapy targeting BCMA;
17. Any conditions judge by investigator for patients not appropriate to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose limitinged toxicity（DLT）after GC012F infusion | Up to 21 days after patients infused with GC012F injectiom
  Incidence of dose-limiting toxicities within 21 days after GC012F infusion.
Adverse Events (AE) after infusion | Up to 48 weeks after patients infused with GC012F injectiom
  Incidence of adverse events within 48 weeks after GC012F infusion

SECONDARY OUTCOMES:
Overall Response Rate(ORR) | Up to 24 weeks after patients infused with GC012F injectiom
  Response assessed according to IMWG criteria (Kumar, Shaji et al. 2016), ORR (sCR, CR,VGPR, and PR) within 24 weeks after infusion Minimal Residual Disease (MRD) assessed by Euroflow ;
Progression-free survival (PFS), Overall Survival (OS), Duration Of Response (DOR) | Up to 1/3/6/9/12 months after patients infused with GC012F injectiom
  Progression-free survival (PFS), overall survival (OS), duration of response (DOR) within 48 weeks after infusion (1/3/6/9/12 months after infusion);
CAR-T cell counts and number of CAR gene copies | Up to 48 weeks after patients infused with GC012F injectiom
  CAR-T cell counts and number of CAR gene copies in the blood, bone marrow and/or tumor tissue within 48 weeks after GC012F infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, MD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China